CLINICAL TRIAL: NCT06341725
Title: Role of Endoscopic Ultrasound to Assess the Lymph Nodes Staging in Non-metastatic Pancreatic Adenocarcinoma
Brief Title: EUS Role in Non-metastatic Pancreatic Adenocarcinoma Lymph Nodes Staging
Status: Terminated | Type: Observational
Why Stopped: no patients with inclusion criteria
Sponsor: Paolo Giorgio Arcidiacono, MD (Other)
Responsible Party: Sponsor-Investigator, Paolo Giorgio Arcidiacono, MD, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: LinfoK EUS 2016
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Adenocarcinoma; Lymph Node Metastasis
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: malignant lymph nodes — observational study

SUMMARY:
Aim of the study will be to investigate if Endoscopic Ultrasound (EUS) with elastography can be purposed between the routine staging examinations in patients with pancreatic adenocarcinoma without distant metastasis for the staging of lymph nodes status ("N" in TNM classification)

* in RESECTABLE pancreatic cancer the investigators will evaluate the concordance with EUS elastography and histological findings of lymph nodes obtained during surgery, in order to assess the sensibility, specificity and the positive and negative predictive value of EUS with elastography, the disease-free survival, the percentage of metastatic patients and the overall survival (in patients with or without metastatic lymph nodes).
* in "BORDERLINE resectable" and UNRESECTABLE non-metastatic ("advanced" locally") disease, the investigators will evaluate if the malignant lymph nodes samples during EUS with elastography and fine needle aspiration (FNA) will be related to a decreased survival.

Secondary aim will be to register the prognosis (in terms of survival) of the patients with para-aortic and mediastinal pathological lymph nodes (related to a decreases survival in some series in literature)

DETAILED DESCRIPTION:
Pathological lymph nodes will be assessed by EUS with elastography as lymph nodes: hypoechoic, rounded, rigid (blue) and big (bigger than 1 centimeter)

ELIGIBILITY:
Inclusion Criteria: pancreatic adenocarcinoma without distant metastasis; patients > 18 years

Exclusion Criteria: distant metastasis and pancreatic adenocarcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pancreatic adenocarcinoma stage I-II and III with malignant lymph nodes assessed by EUS and elastography
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
CONCORDANCE (PERCENTAGE) of pathological lymph nodes at EUS with elastography and surgical pathology report | 2 years
  resectable pancreatic cancer
OVERALL SURVIVAL (MONTHS) in metastatic lymph node presence | 2 years
  resectable pancreatic cancer
OVERALL SURVIVAL (MONTHS) in metastatic lymph node presence | 2 years
  borderline resectable and locally advanced pancreatic cancer

SECONDARY OUTCOMES:
OVERALL SURVIVAL (MONTHS) | 2 years
  para-aortic and mediasitnum metastatic lymph nodes presence

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy